CLINICAL TRIAL: NCT04745221
Title: Efficacy and Safety of Autologous Fecal Bacteria Transplantation in Preventing Acute Graft Versus Host Disease After Haploidentical Hematopoietic Stem Cell Transplantation: a Multicenter, Open, Randomized Controlled Clinical Study
Brief Title: Efficacy and Safety of Auto-FMT in Preventing aGVHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Qi Xiao-Fei, Principal Investigator, The First Affiliated Hospital of Soochow University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FMT2021001
Record Dates: First submitted 2021-02-03; First posted 2021-02-09 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Graft Versus Host Disease, Acute
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- with auto-FMT (Experimental): The patients in the experimental group took autologous fecal bacteria capsule about 3 weeks after bone marrow transplantation.
  Interventions: Other: autologous fecal bacteria
- empty capsule (No Intervention): The patients in this group took empty capsule about 3 weeks after bone marrow transplantation

INTERVENTIONS:
Other: autologous fecal bacteria — autologous fecal bacteria transplantation
  Arms: with auto-FMT

SUMMARY:
To evaluation the efficacy and safety of autologous fecal bacteria transplantation in preventing acute graft versus host disease after haploidentical hematopoietic stem cell transplantation. Bone marrow transplant patients were recruited.

ELIGIBILITY:
Inclusion Criteria:

* Haplo-HSCT patients; Bacteroidetes >0.1%; inverse Simpson diversity ≥2

Exclusion Criteria:

* Gastrointestinal diseases；Age>60; or Age<10；Probiotics or prebiotics were taken before enrollment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Acute Graft-Versus-Host Disease | 90 days after haploidentical hematopoietic stem cell transplantation

SECONDARY OUTCOMES:
overall survival | 90 days after haploidentical hematopoietic stem cell transplantation
Event free survival | 90 days after haploidentical hematopoietic stem cell transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Ye Zhao, Suzhou, Jiangsu, China